CLINICAL TRIAL: NCT03760705
Title: Long-term Clinical Outcomes, Cost-of-care, Clinical Characteristics, Re-admission Rates, Outpatient Care and Mortality in Patients With Coronary Artery Disease or Congestive Heart Failure in Singapore
Brief Title: Singapore Cardiac Longitudinal Outcomes Database
Acronym: SingCLOUD
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Heart Centre Singapore (Other)
Collaborators: Ministry of Health, Singapore (Other Government); Changi General Hospital (Other); National University Hospital, Singapore (Other); Singapore General Hospital (Other); Tan Tock Seng Hospital (Other); Khoo Teck Puat Hospital (Other); SingHealth Polyclinics (Other); National Healthcare Group, Singapore (Other Government); Ng Teng Fong General Hospital (Other); Sengkang General Hospital (Other); National University Polyclinics (Unknown); Alexandra Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CIRB/2013-391/C
Record Dates: First submitted 2018-04-04; First posted 2018-11-30 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2019-12

CONDITIONS: Coronary Artery Disease; Congestive Heart Failure; Atrial Fibrillation
Keywords: CAD; CHF; AF; SingCLOUD; Cardiovascular; Retrospective; BRAIN; HDG; Database
MeSH Terms: conditions — Coronary Artery Disease; Heart Failure; Atrial Fibrillation | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Coronary Artery Disease: 1. Clinical data collected by Singapore Cardiac Data Bank (SCDB)
  2. Clinical, administrative, pharmacy, financial data collected by each participating hospital
  3. Administrative data collected by the Ministry of Health
  Interventions: Other: Data Collection
- Heart Failure: 1. Clinical data collected by Singapore Cardiac Data Bank (SCDB)
  2. Clinical, administrative, pharmacy, financial data collected by each participating hospital
  3. Administrative data collected by the Ministry of Health
  Interventions: Other: Data Collection
- Atrial Fibrillation: 1. Clinical data collected by Singapore Cardiac Data Bank (SCDB)
  2. Clinical, administrative, pharmacy, financial data collected by each participating hospital
  3. Administrative data collected by the Ministry of Health
  Interventions: Other: Data Collection

INTERVENTIONS:
Other: Data Collection — 1. Collection of data as detailed below:
     1. Clinical data collected by SCDB
     2. Clinical, administrative, pharmacy, financial data collected by each participating hospital
     3. Administrative data collected by MOH
  2. Data will be extracted and anonymized on a secure healthcare analytics platform
  3. Collaboration with the MOH for collection of administrative and financial data
  4. Analysis on how healthcare behavior is affected by education, socioeconomic level and other social or cultural factors.
  5. Statistical Analysis by the bio statistical team. This team will be responsible for collecting and merging the collected data and will also ensure the quality of the data.

SUMMARY:
The research project aims to perform data extraction, integration and analysis across multiple clinical, administrative, financial and pharmacy databases in the participating institutions. The key data components will include clinical cardiovascular specific data, procedural data, financial and administrative data (e.g. cost of medications and supplies, length of stay, diagnosis codes etc.), short-to-long term clinical outcomes (including hospital re-admissions, cardiovascular events, death), and quality-of-care indices (e.g. compliance to guideline-recommended therapy and medications). The research project will involve all patients proven and/or suspected with coronary artery disease (CAD), congestive heart failure (CHF) and atrial fibrillation (AF) admitted to National Heart Centre Singapore (NHCS) and NUH.

DETAILED DESCRIPTION:
The research project is initiated by NHCS and its participating institutions include Ministry of Health (MOH), as well as National University Hospital (Singapore) Pte Ltd (NUH), Changi General Hospital (CGH), Khoo Teck Puat Hospital (KTPH), Singapore General Hospital (SGH), Tan Tock Seng Hospital (TTSH), Ng Teng Fong General Hospital (NTFGH) , SingHealth Polyclinics, National Healthcare Group Polyclinics (NHGP), Sengkang Hospital (SKH), National University Polyclinics (NUP), and Alexandra Hospital (AH).

The research project will leverage on the Health Data Grid (HDG) pilot project, now known as Business Research Analytics Insights Network (BRAIN). BRAIN will be a virtual repository that will enable access to anonymised and merged data from disparate databases at multiple institutions. The structures of BRAIN will preserve patients' privacy and confidentiality, ensure IT security and allow access only by authorised persons. The BRAIN pilot project will be co-funded by MOH and the Infocommunication Media Development Authority of Singapore (IMDA). To avoid doubt, after the BRAIN pilot project, a separate approval from the appropriate stakeholders will have to be sought for further funding of the operating costs of the BRAIN, regardless of whether the value of the BRAIN has been demonstrated during the BRAIN pilot project. There is no direct cost involved in the research project.

For the research project, MOH will contribute administrative data from the Registry of Births and Deaths, Casemix & Subvention, the Mediclaim, and Omnibus databases, and the other participating institutions will contribute the data from the National Electronic Health Records (NEHR), Electronic Health Intelligence System (eHIntS) and Enterprise Data Warehouse (EDW) to BRAIN. Only anonymised data from BRAIN will be utilised for the research project.

ELIGIBILITY:
Inclusion Criteria:

* all patients who present to a healthcare institution with either CAD or suspected CAD (including chest pain); CHF or suspected CHF; AF or suspected AF

Exclusion Criteria:

* non-Singaporeans

Ages: 21 Years to 120 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The participating institutions will include National Heart Centre Singapore, National University Heart Centre, Singapore General Hospital, Tan Tock Seng Hospital, Changi General Hospital, Khoo Teck Puat Hospital, Ng Teng Fong General Hospital, Singhealth Polyclinics, National Healthcare Group Polyclinics, Sengkang General Hospital, National University Polyclinics, Alexandra Hospital, and the Ministry of Health Health Services Research Division.
  All patients who present to a healthcare institution with either CAD or suspected CAD (including chest pain); CHF or suspected CHF; AF or suspected AF
Sampling Method: Probability Sample
Enrollment: 7205000 (Estimated)
Dates: Start 2013-07-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure will be to assess the total number of patients who passed away due to any cause at the 1-year time point | 1 year
  Mortality
The primary outcome measure will be to assess the total number of patients who passed away due to any cause at the 2-year time point | 2 year
  Mortality
The primary outcome measure will be to assess the total number of patients who passed away due to any cause at the 3-year time point | 3 year
  Mortality

SECONDARY OUTCOMES:
The secondary outcome measure will be to assess the total number of patients who had major adverse cardiac event (MACE) due to any cause at the 1-year time point | 1 year
  Myocardial Infarction (MI), Stroke, CHF
The secondary outcome measure will be to assess the total number of patients who had MACE due to any cause at the 2-year time point | 2 year
  MI, Stroke, CHF
The secondary outcome measure will be to assess the total number of patients who had MACE due to any cause at the 3-year time point | 3 year
  MI, Stroke, CHF

CONTACTS AND LOCATIONS:
Overall Officials: Khung Keong Yeo, Principal Investigator — National Heart Centre Singapore
Locations (13):
- Singapore (13):
  - National University Hospital (Singapore) Pte Ltd, Singapore
  - National Healthcare Group Polyclinics, Singapore
  - SingHealth Polyclinics, Singapore
  - Alexandra Hospital, Singapore
  - Singapore General Hospital, Singapore
  - National Heart Centre Singapore, Singapore
  - Ministry of Health, Singapore
  - Tan Tock Seng Hospital Pte Ltd, Singapore
  - Changi General Hospital, Singapore
  - National University Polyclinics, Singapore
  - Ng Teng Fong General Hospital, Singapore
  - Khoo Teck Puat Hospital, Singapore
  - Sengkang Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No